CLINICAL TRIAL: NCT03896464
Title: Soft-tissue Quadriceps Autograft ACL-reconstruction in the Skeletally-immature vs. Hamstrings (SQuASH): A Multi-Centre Randomized Controlled Trial
Brief Title: Soft-tissue Quadriceps Autograft ACL-reconstruction in the Skeletally-immature vs. Hamstrings
Acronym: SQuASH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Orthopaedic Foundation (Other); The Physicians' Services Incorporated Foundation (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SQuASH
Record Dates: First submitted 2019-03-27; First posted 2019-04-01 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: ACL - Anterior Cruciate Ligament Rupture
Keywords: Autograft; Soft-tissue hamstring; Quadriceps Tendon
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Autograft donation incisions will be covered with adhesive bandages for clinical outcome assessment by the attending physician. The assessor will perform a physical assessment of the patient's knees, including range of motion and laxity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Soft-tissue hamstring (Active Comparator): All patients in the study will undergo arthroscopic-assisted, single-bundle, complete transphyseal, anatomic primary ACL reconstruction at the discretion of the surgeon, considering the individual patient's age, physeal status, and anticipated years of growth remaining to skeletal maturity. Patients in this arm will undergo soft-tissue autograft reconstruction using hamstrings (i.e. semitendinosus and/or gracilis) grafts. Grafts will be secured on the femur and tibia according to surgeon preference, given literature demonstrating no clear superior method for graft fixation.
  Interventions: Procedure: Soft tissue hamstring autograft
- Quadriceps tendon (Active Comparator): Patients in this arm will undergo soft-tissue autograft reconstruction using all-soft-tissue quadriceps (i.e. full or partial thickness) grafts. Grafts will be secured on the femur and tibia according to surgeon preference, given literature demonstrating no clear superior method for graft fixation.
  Interventions: Procedure: Quadriceps tendon autograft

INTERVENTIONS:
Procedure: Soft tissue hamstring autograft — Patients will be prescribed to receive a soft tissue hamstring autograft to for ACL reconstruction.
  Arms: Soft-tissue hamstring
Procedure: Quadriceps tendon autograft — Patients will be prescribed to receive a quadriceps tendon autograft to for ACL reconstruction.
  Arms: Quadriceps tendon

SUMMARY:
To date, the use of the quadriceps tendon as an autograft option in primary paediatric Anterior Cruciate Ligament (ACL) reconstruction has not been well studied. The 2018 International Olympic Committee (IOC) Consensus Statement now outlines the quadriceps tendon as a possible autograft option. However, no Randomised Control Trial (RCT) has examined the efficacy of the quadriceps tendon autograft in primary paediatric ACL reconstruction compared to the historical "gold-standard" soft-tissue hamstring autograft in this population. In light of its evidence for favourable outcomes in the adult population, and the (albeit limited) evidence showing safety and promise in the paediatric population, clinical equipoise exists for assessing its impact on outcomes in paediatric patients at the index surgery. This is a parallel, international, multi-centre, blinded randomized controlled trial of 352 skeletally-immature (at the time of injury) patients (ages 10-18 years, inclusive) undergoing primary ACL reconstruction to compare the effect of autograft tendon choice (i.e. hamstring versus soft-tissue quadriceps) on the rates of ACL graft failure, return-to-sport, knee function, pain, health-related quality of life and health utility, psychological factors, range of motion and stability, and any other adverse events at 24 months.

ELIGIBILITY:
Inclusion Criteria

1. Patients aged 10-18 years.
2. History, physical exam, and magnetic resonance imaging (MRI) or arthroscopic image confirmation of ACL insufficiency.
3. Suitable for anatomic, single-bundle arthroscopic-assisted ACL reconstruction.
4. X-ray or MRI evidence of skeletal immaturity (i.e., open physes) based on imaging that is closest to the time of injury (and correlated with standard bone age left hand posteroanterior (PA) radiographs).
5. Patient involved in sport (competitive and/or recreational level) prior to injury.
6. Patient and parent/guardian speak, read, and understand the language of the clinical site.
7. Patient and parent/guardian provide informed consent and/or assent.

Exclusion Criteria

1. Evidence (i.e. radiographic and/or arthroscopic) of International Cartilage Repair Society (ICRS) Cartilage Lesion Classification System Grade 2 (i.e., lesions extending down to 50% of the cartilage depth) and higher osteoarthritis that is symptomatic, requiring treatment other than debridement or microfracture.
2. Tibial eminence/spine fractures treated surgically.
3. Concomitant collateral, posterior cruciate, and/or cartilage pathology requiring surgical reconstruction and/or advanced restoration techniques (i.e., osteochondral allograft or autograft transfer, matrix-induced autologous chondrocyte implantation, particulate juvenile articular cartilage allograft transplantation).
4. Previous ACL reconstruction in the affected knee or contralateral knee.
5. Previous distal femur and/or proximal tibial/fibular physeal injury in the affected knee or contralateral knee.
6. Allograft or allograft-augmentation, or synthetic augmentation of the ACL reconstruction.
7. Biological-augmentation of the ACL reconstruction (i.e. platelet-rich-plasma, fibrin clot, reinforced bioinductive implants, etc.).
8. ACL reconstruction utilizing synthetic grafts.
9. Primary ACL repair.
10. Patient diagnosed with inflammatory arthropathy.
11. Significant medical co-morbidities (requiring daily assistance for activities of daily living).
12. Patient, parent/guardian, and/or clinical investigator believe the patient will have difficulty maintaining follow-up.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 352 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Rate of ACL failure | 2 years
  ACL graft failure is a composite outcome defined by MRI confirmation of rupture and/or asymmetrical symptomatic laxity (i.e., positive Lachman and/or positive pivot shift).

SECONDARY OUTCOMES:
Rate of Return to Sport | 2 years
  Return to sport (at any level and to pre-injury level) will be evaluated using the Tegner Activity Scale. The Tegner activity level scale is a graduated list of activities of daily living, recreation, and competitive sports, in which the response is presented as an 11-point Likert scale, where 0 indicates the lowest level of ability to perform work and sport functions, and 10 indicates competitive participation in high level sports.
Patient Reported Knee Function | 2 years
  Patient Knee Function will be evaluated using the Pediatric International Knee Documentation Committee Subjective Form (Pedi-IKDC). The Pedi-IKDC is a 15 question form that consists of measures of daily living and sport activity, in which the response options are presented as either 4 or 10 point Likert scales. Scores for the form range from 0 (lowest level of function) to 100 (highest level of function).
Knee Pain | 2 years
  Knee pain will be evaluated using a 100-point Visual Analogue Scale (VAS). The VAS has been validated in ACL patients and is one of the most commonly used pain rating scores both in research and clinical practice as it is an easy-to-use, validated, one-dimensional scale that does not require verbal or reading skills.
Health-Related Quality of Life | 2 years
  Health-related quality of life (HRQL) and health utility will be evaluated using the EuroQol 5 Dimensions for Youth (EQ-5D-Y-3L) questionnaire.The EQ-5D is a standardized, utility-based instrument for use as a measure of HRQL and health utility. Similar to the adult version, the EQ-5D-Y-3L comprises 5 questions on mobility, self-care, usual activities, pain/discomfort, and anxiety/ depression. The EQ-5D-Y-3L has been extensively validated in international paediatric populations.
Psychological Readiness to Return-to-Sport | 2 years
  Psychological predictors, specifically psychological readiness to return-to-sport, will be evaluated using the Anterior Cruciate Ligament Return to Sport after Injury (ACL-RSI) questionnaire, which has been shown to be reliable and responsive at the group (study) level in younger populations across all sexes. The ACL-RSI scale has 3 domains: risk appraisal, confidence, and emotions. Greater psychological preparation is indicated by higher scores.
Range of Motion | 2 years
  Knee range of motion (ROM) and both anterior-posterior and rotational stability will be evaluated through physical examination (i.e. Lachman and pivot shift tests, respectively). ROM will be measured in the flexion-extension (i.e. sagittal) plane using a goniometer. Anterior-posterior stability will be measured using the Lachman test, given its non-invasive nature, high sensitivity, superiority over the anterior drawer test, and by virtue of being the most reliable clinical method to assess ACL integrity. It will be performed in the supine position, with the extremity in 20-30° of knee flexion, as is commonly described. Similarly, rotational stability will be assessed using the standardized pivot shift test, performed in 30° of knee flexion.
Adverse Events | 2 years
  The expert Adjudication Committee will evaluate all graft failures, re-operations and other knee-related adverse events through a process of independent review and consensus, guided by decision rules detailed in the Adjudication Charter (drafted using recommendations from the literature, tested for validity and agreement among the adjudicators, and in use for the pilot study). An adverse event is defined as any symptom, sign, illness, or experience that develops or worsens in severity during the course of the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Darren de SA, MD, FRCSC, Principal Investigator — McMaster University
Locations (6):
- Canada (5):
  - McMaster University, Hamilton, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Women's College Hospital/Research Institute, Toronto, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
  - Shriners Hospitals for Children - Canada, Montreal, Quebec
- Kobe University, Kobe, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ayeni OR; SQuASH Investigators. Soft-tissue quadriceps tendon autograft during primary anterior cruciate ligament reconstruction in Skeletally-immature patients vs. Hamstrings: A protocol for a multi-centre randomized controlled trial. J Orthop Surg Res. 2025 Dec 1;21(1):6. doi: 10.1186/s13018-025-06534-0. PMID 41327264